CLINICAL TRIAL: NCT07251127
Title: A Single-dose, Randomized, Crossover, Comparative Bioavailability Study of 500 mg Metronidazole Delayed-release (DR) Capsules of Gateway Pharmaceutical LLC, USA and Metronidazole Tablets USP in Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Study of Metronidazole Delayed-Release Capsules in Comparison With Immediate-Release Tablets (Flagyl) for Safety and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gateway Pharmaceutical LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP-MTZ DR-25-0527
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Clostridium Difficile Infection (CDI)
Keywords: Metronidazole; Delayed-release; Phase 1; Pharmacokinetic; Clostridium difficile infection; Colon-targeting; Colon-delivery; 505b2
MeSH Terms: conditions — Clostridium Infections | interventions — Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metronidazole DR Capsule (Experimental): Colon-delivery
  Interventions: Drug: Delayed-release metronidazole
- Metronidazole Tablet USP (Active Comparator): Immediate-release
  Interventions: Drug: Immediate-release metronidazole

INTERVENTIONS:
Drug: Delayed-release metronidazole — Oral single dose, 500 mg
  Other Names: 505(b)(2)
  Arms: Metronidazole DR Capsule
Drug: Immediate-release metronidazole — Oral single dose, 500 mg
  Other Names: Flagyl®
  Arms: Metronidazole Tablet USP

SUMMARY:
Clostridium difficile Infection (CDI) also referred to as Clostridium difficile associated diarrhea (CDAD) is an infectious disease that is commonly associated with taking broad-spectrum antimicrobials and certain cancer chemotherapy drugs, which unbalance the ecosystem of the colon causing Clostridium difficile to become the predominant part of the microbiota. C. difficile is a Gram-positive anaerobe, non-invasive by remaining in the colon lumen, and produces toxins A and B that cause diseases, ranging from diarrhea, to pseudomembranous colitis, toxic megacolon, colon perforation, sepsis, or death.

CDI is the leading cause of hospital-associated gastrointestinal illness, responsible for ~ 500,000 infections and 29,000 deaths each year in the US. It places a high burden on the health-care system, which costs $4.8 billion annually. Rates of CDI have been increasing since 2000, especially in the elderly with a recent hospitalization or residing in long-term care facility (LTCF). The mortality rate from CDI is 2 to 5% but increases to 10 to 20% among elderly debilitated patients, and is even greater in patients who develop severe colitis or systemic toxicity. More recently, it has become a community pathogen, affecting younger populations who were previously at low risk.

Currently there are limited medicines for treating active CDI, and no new antibiotic approvals in this area after 2011. Fidaxomicin is concerned with its cost and increased burden of resistance; Vancomycin is related to vancomycin-resistant enterococci and saved as the last resort antibiotic; metronidazole as immediate-release tablets (Flagyl) is completely absorbed from the upper GI tract into the systemic blood systems, leaving low and inconsistent drug concentrations at the colon to battle C. difficile. More treatment options are urgently needed.

Gateway Pharma has developed a 505(b)(2) new product, Metronidazole Delayed-Release (DR) Minitablets in Capsule using our patent-protected colon-targeting platform. The goal is to reduce metronidazole blood absorption and increase drug local concentrations at the colon, to achieve 1) improved efficacy and 2) reduced side effects. Our ultimate goal is to restore metronidazole as the first-line medicine for treating CDI.

DETAILED DESCRIPTION:
To compare the absorption rate and extent of the DR Capsule with the IR Tablet, to measure the amount of metronidazole in feces and to monitor the safety and tolerability of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 45 years (both inclusive).
2. Subjects' weight within normal range according to normal values for Body Mass Index (between 18.5 and 30.0 kg/m2) (both inclusive) with minimum of 45 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the normal range.
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. Subjects having normal chest X-Ray (PA view), if taken.
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Subjects having negative urine alcohol test / breath alcohol test.
8. Non-smoker.
9. Subjects willing to adhere to the protocol requirements and to provide written informed consent.
10. Subjects having negative urine pregnancy test at screening and negative serum b-hCG pregnancy test on admission day of period 01 (only for female subjects).

Exclusion Criteria:

1. Hypersensitivity to Metronidazole, nitroimidazole derivatives or related class of drugs or any of its excipients or heparin.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, urogenital or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 30 days prior to admission in period 01.
4. Presence of alcoholism or drug abuse.
5. History or presence of asthma, urticaria or other significant allergic reactions.
6. Subjects with known history of Cockayne's syndrome
7. History or presence of significant gastric and/or duodenal ulceration.
8. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
9. History or presence of cancer or basal or squamous cell carcinoma.
10. Consumption of xanthine-containing products, tobacco containing products or alcohol or any alcohol containing products within 48.00 hours prior to admission in period 01.
11. Consumption of grapefruit or grapefruit juice containing products within 72.00 hours prior to admission of period 01.
12. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
13. History or presence of significant easy bruising or bleeding.
14. History or presence of significant recent trauma.
15. Female subjects who are currently breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve | up to 3 days
Cmax | up to 3 days

SECONDARY OUTCOMES:
Occurrence of adverse events | up to 7 days
Fecal drug level | up to 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Veeda Lifesciences, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grundfest-Broniatowski S, Quader M, Alexander F, Walsh RM, Lavery I, Milsom J. Clostridium difficile colitis in the critically ill. Dis Colon Rectum. 1996 Jun;39(6):619-23. doi: 10.1007/BF02056938. PMID 8646945
- [Result] Debast SB, Bauer MP, Kuijper EJ; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases: update of the treatment guidance document for Clostridium difficile infection. Clin Microbiol Infect. 2014 Mar;20 Suppl 2:1-26. doi: 10.1111/1469-0691.12418. PMID 24118601
- [Result] Cohen SH, Gerding DN, Johnson S, Kelly CP, Loo VG, McDonald LC, Pepin J, Wilcox MH; Society for Healthcare Epidemiology of America; Infectious Diseases Society of America. Clinical practice guidelines for Clostridium difficile infection in adults: 2010 update by the society for healthcare epidemiology of America (SHEA) and the infectious diseases society of America (IDSA). Infect Control Hosp Epidemiol. 2010 May;31(5):431-55. doi: 10.1086/651706. PMID 20307191